CLINICAL TRIAL: NCT03186053
Title: Cardioprotective Effects of Sodium Creatine Phosphate in Valve Surgery: A Prospective Randomized Controlled Study
Brief Title: Sodium Creatine Phosphate in Heart Valve Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Guyan Wang, The Chief of Infection-Control Department, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FWT2017-ZX004
Record Dates: First submitted 2017-05-29; First posted 2017-06-14 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases | interventions — Phosphocreatine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium creatine phosphate (Experimental): 5g creatine phosphate was dissolved in 50ml saline solution. After induction of anesthesia, the patients were first given a load dose of 1g, 20min (30ml / h) , And then pumped at a rate of 1 g / h (10 ml / h).
  Interventions: Drug: sodium creatine phosphate
- Control (Placebo Comparator): The control group was treated with saline in the same manner.
  Interventions: Drug: saline

INTERVENTIONS:
Drug: sodium creatine phosphate — sodium creatine phosphate .Loading dose followed by continuous infusion in operation
  Other Names: Neoton
  Arms: sodium creatine phosphate
Drug: saline — .Loading dose followed by continuous infusion in operation
  Arms: Control

SUMMARY:
To explore the effect of intraoperative sodium creatine phosphate on myocardial protection in patients undergoing valve surgery

DETAILED DESCRIPTION:
Objective: To explore the effect of intraoperative sodium creatine phosphate on myocardial protection in patients undergoing valve surgery Methods: 250 patients undergoing valve surgery were randomly divided into experimental group and control group. 5g creatine phosphate was dissolved in 50ml saline solution. After induction of anesthesia, the patients were first given a load dose of 1g, 20min (30ml / h) , And then pumped at a rate of 1 g / h (10 ml / h). The control group was treated with saline in the same manner. The cTnI level was measured at the corresponding time points. Hemodynamic indexes and postoperative complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* valvular disease patients requiring valvular replacement or repair surgery with cardiopulmonary bypass(CPB)

Exclusion Criteria:

* thoracoscopic valve surgery
* other organ dysfunction: such as cancer, organ failure, severe anemia, infection
* patients with mental disorders
* coagulopathy, active ulcer, ischemic or hemorrhagic stroke (within 6 months), trauma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
serum cardiac troponin I(cTnI) | within 24 hours after aortic declamping
  serum cardiac troponin I(cTnI)

SECONDARY OUTCOMES:
mortality | within 30 postoperative days
  death rate in hospital
stroke | within 30 postoperative days
  defintion by surgeon
blood filtration of kidney failure | within 30 postoperative days
  need for dialysis
extracorporeal membrane oxygenation (ECMO) or intraaortic balloon counterpulsation (IABP) support | within 30 postoperative days
  heart failure requires mechanical assistance
mechanical ventilation time | within 30 postoperative days
  ventilation
arrhythmia | within 30 postoperative days
  Atrial fibrillation or Ventricular fibrillation or Ventricular tachycardia requiring drug treatments

CONTACTS AND LOCATIONS:
Overall Officials: Guyan WANG, M.D., Study Director — Department of anesthesiology,Fuwai hospital
Locations (2):
- China (2):
  - Department of Anesthesiology ,Fuwai Hospital, National Center for Cardiovascular Diseases, CAMS and PUMC, Beijing, Beijing Municipality
  - Cardiovascular Institute and Fuwai Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No